CLINICAL TRIAL: NCT01518335
Title: A Double-Blind, Randomized, Placebo Controlled Study Evaluating the Use of Platelet Rich Plasma Therapy for Acute Ankle Sprains in the Emergency Department.
Brief Title: Use of Platelet Rich Plasma Therapy for Acute Ankle Sprains in the Emergency Department
Acronym: PRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein Healthcare Network (Other)
Responsible Party: Principal Investigator, James Gardner, MD, MD, Albert Einstein Healthcare Network
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HN4157
Record Dates: First submitted 2011-12-08; First posted 2012-01-26 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Sprain of Ankle
Keywords: platelet rich plasma; ankle; sprain; injection; Platelet Rich Plasma therapy; focal, invasive therapy for sprains
MeSH Terms: conditions — Ankle Injuries; Sprains and Strains | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Platelet Rich Plasma (Experimental): Patients receive Platelet rich plasma injection + standard of care therapy(bandaging or boot and crutches) + non-NSAID pain medicine
  Interventions: Procedure: Platelet rich plasma injection
- Placebo/Standard of Care (Placebo Comparator): Patient receives Placebo Comparator: Placebo/Standard of Care [saline injection + standard of care (bandaging or boot and crutches)] + non-NSAID pain medicine
  Interventions: Procedure: Placebo Comparator: Placebo/Standard of Care

INTERVENTIONS:
Procedure: Platelet rich plasma injection — 50ml of blood drawn into a 60cc with 10cc of anticoagulant is processed using MAGELLAN® Autologous Platelet (Arteriocyte Medical Systems, Cleveland Ohio)to separate out approximately 3-6 cc of platelet rich plasma, which is mixed with 1 cc of 1 % Lidocaine (xylocaine) and 1 cc of 0.25 % Marcaine (bupivacaine) and injected into the site of injury under USG guidance.
  Arms: Platelet Rich Plasma
Procedure: Placebo Comparator: Placebo/Standard of Care — 50ml of blood is drawn into a 60cc with 10cc of anticoagulant and is then discarded. 4 cc of saline solution is mixed with 1 cc of 1 % Lidocaine (xylocaine) and 1 cc of 0.25 % Marcaine (bupivacaine) and injected into the site of injury under USG guidance.
  Arms: Placebo/Standard of Care

SUMMARY:
This research study hopes to determine whether or not platelet rich plasma therapy improves healing time of moderate to severe ankle sprain in comparison to standard of care therapy.

DETAILED DESCRIPTION:
The intention of this research project is to study a new treatment for severe ankle sprains.This new treatment is called Platelet Rich Plasma (PRP) therapy and involves injecting concentrated platelet's from a patient's own blood into the site of injury to aid healing. Platelets, aside from their clotting capabilities also serve a role in re-vascularization of tissue as well as collagen repair. PRP therapy has been used in sports medicine for treatment of chronic injuries but has yet to be proven effective in acute injury of a joint. The investigators are comparing treatment and placebo groups based on a subjective patient questionnaire and pain score administered on the day of injury and 2-3 days and 8-10 days follow up.

ELIGIBILITY:
Inclusion Criteria:

* severe ankle sprain
* X-ray completed

Exclusion Criteria:

* Pregnancy/breastfeeding
* Police custody
* active infection
* metastatic disease/tumors
* History of thrombocytopenia
* Allergy to ester or amine anesthetics
* On anticoagulant medication
* Peripheral vascular disease
* Known coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-06; Primary Completion 2012-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline of LEFS score, a previous validated 80-point scale used to quantify lower extremity function. | Day 0; Day2-3; Day 8-10; Day30
  The primary outcome of this investigation is change from baseline in LEFS score, a previous validated 80-point scale used to quantify lower extremity function. A difference of 9 points is considered clinically significant.

SECONDARY OUTCOMES:
Change in pain from baseline | Day 0; Day 2-3, Day 8-10, Day 30
  Changes in level of pain from baseline was measured using VAS scale as well as comparing need for narcotics use at each follow up time point.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Rowden, DO, Principal Investigator — Eisntein Healthcare Network
Locations (1):
- Einstein Healthcare Network, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No